CLINICAL TRIAL: NCT07172802
Title: An Open-label, Multicenter, Dose Escalation and Expansion Phase 1/2 Study to Evaluate the Safety, Tolerability and Pharmacokinetics, and Anti-tumor Activity of GI-108, an Anti-CD73-IgG4 Fc-IL-2v Bispecific Fusion Protein, as a Single Agent in Patients With Advanced or Metastatic Solid Tumors
Brief Title: A Study of GI-108, an Anti-CD73-IgG4 Fc-IL-2v Bispecific Fusion Protein, as Monotherapy in Patients With Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GI Innovation, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GII-108-P101
Record Dates: First submitted 2025-08-28; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Advanced Solid Tumor; Metastatic Solid Tumor; Non-small Cell Lung Cancer (NSCLC); Head and Neck (HNSCC); Pancreatic Cancer; Renal Cell Carcinoma (RCC)
Keywords: GI-108
MeSH Terms: conditions — Neoplasm Metastasis; Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck; Pancreatic Neoplasms; Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GI-108 (Experimental): Dose escalation: GI-108 intravenous (IV), multiple ascending doses Dose optimization: GI-108 intravenous (IV), sRP2D
  Interventions: Drug: GI-108

INTERVENTIONS:
Drug: GI-108 — Dose level will be escalated from 0.1mg/kg to 0.6 mg/kg and Recommended phase 2 dose (or RP2D) of GI-108 will be administered via IV infusion Q3W upto 2 years (approximately 35 years)

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics, and therapeutic activity of GI-108, as a single agent, in patients with advanced or metastatic solid tumors

DETAILED DESCRIPTION:
This is an open-label, multicenter, dose escalation and expansion, phase 1/2 study to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD) and anti-tumor activity of GI-108 as a single agent in advanced or metastatic solid tumors. A control arm is not included.

The study is composed of two phases:

* Dose escalation phase
* Dose expansion phase The dose escalation phase will enroll up to 36 patients with advanced or metastatic solid tumors. At least 3 dose-limiting toxicity (DLT) evaluable patients will be enrolled in each cohort during the dose escalation to establish a maximum tolerated dose (MTD) or tentative recommended phase 2 dose (RP2D). Enrollment in each cohort may be extended to enroll additional 4~7 patients (aiming to recruit upto 10 patients including DLT evaluable patients per cohort), potentially enriched in certain tumor types and/or characteristics to confirm safety, PK and/or pharmacodynamics (PD) of GI-108. The Safety Monitoring Committee (SMC) will determine extension of each cohort based on the review of all available clinical data including efficacy, safety, PK and/or PD. Of the 4 planned cohorts in the dose escalation phase, up to 3 cohorts may be extended to include additional patients based on safety, efficacy PK and/or PD data. The evidence of enrollment extension should be documented for each cohort during dose escalation phase.

ELIGIBILITY:
Key Inclusion Criteria:

* Males and females aged ≥ 18 years (or ≥ 19 years according to local regulatoryguidelines) at the time of screening.
* Has adequate organ and marrow function as defined in protocol.
* Measurable disease as per RECIST v1.1.
* ECOG performance status 0-1.
* Adverse events related to any prior chemotherapy, radiotherapy, immunotherapy,other prior systemic anti-cancer therapy, or surgery must have resolved to Grade≤1, except alopecia and Grade 2 peripheral neuropathy.
* HIV infected patients must be on anti-retroviral therapy (ART) and have a well-controlled HIV infection/disease as defined in protocol.

Key Exclusion Criteria:

* Has known active CNS metastases and/or carcinomatous meningitis. An active second malignancy.
* Has active or a known history of Hepatitis B or known active Hepatitis C virus infection.
* Has active tuberculosis or has a known history of active tuberculosis. Active or uncontrolled infections, or severe infection within 4 weeks before study treatment administration.
* History of chronic liver disease or evidence of hepatic cirrhosis, except patients with liver metastasis.
* Has an active autoimmune disease that has required systemic treatment in past 2 years.
* Previous immunotherapies related to mode of action of GI-102. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroidtherapy or any other form of immunosuppressive medications within 2 weeksprior to Cycle 1 Day 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose-Limiting Toxicities (DLTs) (Dose escalation phase) | Study Day 1, assessed up to DLT period (3 weeks after treatment)
  Number and proportion of subjects experiencing DLTs during dose escalation, used to determine MTD and/or RP2D.
Incidence and Severity of Immune-Related Adverse Events (irAEs) (Dose escalation phase) | From Day 1 through study completion (up to ~24 months)
  Number and proportion of subjects with immune-related AEs, graded per CTCAE v5.0.
Objective Response Rate (ORR) according to RECIST version 1.1 (Dose expansion phase) | Study Day 1, assessed up to approximately 24 months
  Based on Investigator review of radiographic imaging

SECONDARY OUTCOMES:
Objective Response Rate (ORR) according to RECIST version 1.1 (Dose escalation phase) | Study Day 1, assessed up to approximately 24 months
  Based on Investigator review of radiographic imaging
Incidence and Severity of Immune-Related Adverse Events (irAEs) (Dose expansion phase) | Day 1 through study completion, up to ~24 months
  Number and proportion of subjects with immune-related AEs, graded per CTCAE v5.0.
Disease Control Rate (DCR) | Study Day 1, assessed up to approximately 24 months
  DCR is defined as the percentage of patients who have achieved CR, PR and stable disease (SD), per RECIST v1.1 guideline as determined by the investigators.
Duration of objective response (DoR) | Study Day 1, assessed up to approximately 24 months
  DCR is defined as the time from the first occurrence of a documented objective response to the time of the first document disease progression or death from any cause, whichever occurs first, per RECIST v1.1 as determined by the investigator.
Progression-free survival (PFS) | 6-month, 12-month, and 18-month
  PFS is defined as the time from the first study treatment (Day 1) to the first occurrence of progression or death from any cause, whichever occurs first, per RECIST v1.1 guideline as determined by the investigator
Overall survival (OS) | 12-month and 18-month
  OS is defined as the time from the first study treatment to death from any cause
Peak plasma concentration (Cmax) of GI-108 | Study Day 1, assessed up to approximately 24 months
  Based on the concentration vs time profile by dose level
Half-life of GI-108 (T1/2) | Study Day 1, assessed up to approximately 24 months
  Based on the concentration vs time profile by dose level
Area under the plasma concentration versus time curve (AUC) of GI-108 | Study Day 1, assessed up to approximately 24 months
  Based on the concentration vs time profile by dose level
Clearance of GI-108 | Study Day 1, assessed up to approximately 24 months
  Based on the concentration vs time profile by dose level
Volume of distribution (Vd) of GI-108 after administration | Study Day 1, assessed up to approximately 24 months
  Based on the concentration vs time profile by dose level

OTHER OUTCOMES:
Immunophenotyping of peripheral blood mononuclear cells | Study Day 1, assessed up to approximately 24 months
  Peripheral immune cell subpopulation (e.g., CD4+ T cells, CD8+ T cells, regulatory T cells) will be assessed.
Incidence of anti-GI-102 antibody (ADA) and neutralizing antibody (Nab) | Study Day 1, assessed up to approximately 24 months
  Serum will be assessed for the presence of ADA and Nab based on the appropriate assay.

CONTACTS AND LOCATIONS:
Locations (3):
- South Korea (3):
  - Yonsei University Health System, Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No